CLINICAL TRIAL: NCT03113201
Title: Projekt Collabri Flex - The Effect of a Danish Model for Collaborative Care for People With Depression in General Practice
Brief Title: Collabri Flex - Effect of Collaborative Care for People With Depression in General Practice
Acronym: Collabri Flex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amager Hospital (Other)
Responsible Party: Principal Investigator, Lene Falgaard Eplov, Head of Research, Associate professor, Amager Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Collabri Flex - Depression
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Depression
Keywords: Depression; Collaborative care; Care manager; Anxiety; Psychiatry; Consultation-liaison; General practitioner
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collabri Flex (Experimental): Collaborative care
  Interventions: Behavioral: Collaborative care
- Consultation-Liaison (Experimental): Consultations with general practitioner
  Interventions: Behavioral: Consultations-Liaison

INTERVENTIONS:
Behavioral: Collaborative care — Collaborative care provided by the general practitioner and the care manager. Treatment modalities: Cognitive-behavior Therapy, psychoeducation and medication according to a stepped care model
  Arms: Collabri Flex
Behavioral: Consultations-Liaison — Consultation-Liaison provided by general practitioner involving a educational relationship with the Collabri Flex team (care manager and psychiatrist).
  Arms: Consultation-Liaison

SUMMARY:
The aim of the study Collabri Flex is to:

* Develop a Danish model for collaborative care for patients with depression in general practice, based on past experience gained in the Collabri Project.
* Examine the impact of this model compared with liaison-consultation for people with depression in a randomized controlled design from selected endpoints.

DETAILED DESCRIPTION:
The Collabri Flex model for Collaborative Care takes point of departure in the earlier study Collabri. It is changed according to gathered information under the first study of the Collabri model in order to achieve a Danish Collaborative Care model easier to implement.

The aims of Project Collabri Flex are to:

* Develop a flexible model for collaborative care (the Collabri Flex model) for patients with depression.
* Study the effects of this Collabri Flex model against consultation liaison in a randomized design on selected outcomes.

In Collabri the treatment is in line with a set of general treatment principles relevant for collaborative care interventions. The patients in the intervention group are offered cognitive behavioral therapy (CBT), psychoeducation and medication according to a stepped care model by a care manager refering to the general practitioner.

The Collabri Flex study is set up as a researcher-blinded individually randomized controlled trial with participation of an intervention group (treatment according to the Collabri Flex model) and a consultation liaison group.

This study will contribute with new knowledge on collaborative care interventions in a Scandinavian context.

ELIGIBILITY:
Inclusion Criteria:

* Danish speaking
* Diagnosis of current depression based on the Mini International Neuropsychiatric Interview (MINI) by care managers that have been trained in using MINI in close collaboration with the psychiatrist/psychologist.
* The patient has given her/his written informed consent to participate in the trial at the described terms

Exclusion Criteria:

* High risk of suicide assessed in the Mini International Neuropsychiatric Interview (MINI) and/or by the GP
* Psychotic condition detected in the MINI and/or by the GP
* Patients with a diagnosis of dementia
* Alcohol or substance misuse that hinders the person participating in Collabri treat-ment as assessed by the practitioner or care manager at inclusion interview
* If the patient has been referred or is recommended referral to secondary care treatment (mental health center) or psychiatrist in private practice
* Patients who are assessed by the GP as medically unstable making it impossible for the patient to adhere to treatment
* Bipolar affective disorder as assessed in the MINI and/or by the GP
* Pregnancy

For patients in the Collabri Flex group:

* Patients with depression who wants treatment cf. the psychologist scheme (Psykologordningen) or similar treatment and do not want the refferal to the psychologist preceded by other treatment, cf. the Collabri Flex model assessed by the GP
* Patients that wish to continue current psychological or psychiatric treatment due to anxiety or depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Self-reported degree of depression | 6 months
  Measured by Beck Depression Inventory (BDI-II)

SECONDARY OUTCOMES:
Self-reported degree of anxiety | 6 months
  Measured by Beck anxiety Inventory (BAI)
Self-reported psychological stress | 6 months
  Measured by Symptom Checklist (SCL-90-R)
Self-reported functional impairment | 6 months
  Measured by Sheehan disability Scale (SDS)
Self-reported quality of life/well-being | 6 months
  Measured by WHO-5

OTHER OUTCOMES:
Sick leave | 6 months
  Obtained from the DREAM database
Sick leave | 18 months
  Obtained from the DREAM database
Self-reported self-efficacy | 6 months
  Measured by personal control (IPQ-R scale) and two subscales from the Chronic Disease Self-Efficacy Scales; Obtain help from Comunity, Family, Friends Scale and Control/manage Depression Scale
Self-reported self-efficacy | 18 months
  Measured by personal control (IPQ-R scale) and two subscales from the Chronic Disease Self-Efficacy Scales; Obtain help from Comunity, Family, Friends Scale and Control/manage Depression Scale
Self-reported health-related quality of life | 6 months
  Measured by EQ-5D
Self-reported health-related quality of life | 18 months
  Measured by EQ-5D
Self-reported experience of support in recovery | 6 months
  Experience of support in recovery (INSPIRE)
Employment | 6 months
  Obtained from the DREAM database
Employment | 18 months
  Obtained from the DREAM database
Mental-health outpatient services | 6 months
  Obtained from LPR
Mental-health outpatient services | 18 months
  Obtained from LPR
Patient satisfaction | 6 months
  Self-reported experience of satisfaction with treatment (CSQ-8)
Self-reported degree of depression | 18 months
  Measured by Beck Depression Inventory (BDI-II)
Self-reported degree of anxiety | 18 months
  Measured by Beck anxiety Inventory (BAI)
Self-reported psychological stress | 18 months
  Measured by Symptom Checklist (SCL-90-R)
Self-reported functional impairment | 18 months
  Measured by Sheehan disability Scale (SDS)
Self-reported quality of life/well-being | 18 months
  Measured by WHO-5

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Eplov, MD, PhD, Principal Investigator — Research Unit, Mental Health Center Copenhagen
Locations (1):
- Mental Health Centre Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Curth NK, Bjorkedal STB, Hjorthoj C, Brinck-Claussen U, Jorgensen KB, Rosendal S, Bojesen AB, Nordentoft M, Eplov LF. Collaborative Care Versus Consultation Liaison for Patients With Depression or Anxiety Disorders in General Practice in Denmark: 18-Month Follow-Up From the Collabri Flex Trials. Depress Anxiety. 2025 Jun 5;2025:2909617. doi: 10.1155/da/2909617. eCollection 2025. PMID 40510804
- [Derived] Curth NK, Hjorthoj C, Brinck-Claussen U, Jorgensen KB, Rosendal S, Bojesen AB, Nordentoft M, Eplov LF. The effects of collaborative care versus consultation liaison for anxiety disorders and depression in Denmark: two randomised controlled trials. Br J Psychiatry. 2023 Sep;223(3):430-437. doi: 10.1192/bjp.2023.77. PMID 37395101
- [Derived] Curth NK, Brinck-Claussen U, Jorgensen KB, Rosendal S, Hjorthoj C, Nordentoft M, Eplov LF. Collaborative care vs consultation liaison for depression and anxiety disorders in general practice: study protocol for two randomized controlled trials (the Danish Collabri Flex trials). Trials. 2019 Oct 25;20(1):607. doi: 10.1186/s13063-019-3657-0. PMID 31653228